CLINICAL TRIAL: NCT01065532
Title: Healing Responses After Treatment of Bare Metal Stent Restenosis With Implantation of an Everolimus-eluting Xience V Stent Versus Use of a Paclitaxel-eluting Balloon: Optical Coherence Tomography Study
Brief Title: SEDUCE OCT Study in Coronary Artery rEstenosis:an Optical Coherence Tomography (OCT) Study
Acronym: SEDUCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2009-011440-20
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2018-10

CONDITIONS: Restenosis
Keywords: Restenosis; PCI; Drug-eluting stent; Drug-eluting balloon; Optical Coherence Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): SeQuent Please Drug-eluting balloon
  Interventions: Device: Sequent Please Paclitaxel eluting balloon
- 2 (Active Comparator): Xience V Drug-eluting stent
  Interventions: Device: Xience V everolimus eluting stent

INTERVENTIONS:
Device: Sequent Please Paclitaxel eluting balloon — Sequent Please Paclitaxel eluting balloon
  Arms: 1
Device: Xience V everolimus eluting stent — Xience V everolimus eluting stent
  Arms: 2

SUMMARY:
Different healing responses after treatment of bare metal stent restenosis with implantation of an everolimus-eluting Xience V stent (Abbott Vascular) versus use of a paclitaxel-eluting SeQuent Please balloon (BBraun): an optical coherence tomography study.

A prospective, single-centre, randomized clinical trial with clinical, angiographic and OCT follow-up at 9 months.

DETAILED DESCRIPTION:
Background: The optimal treatment of bare metal stent restenosis (implantation of a drug-eluting stent, simple balloon dilatation, CABG) is still not defined. The most used option nowadays is the implantation of a drug-eluting stent (DES). However, this procedure implies application of a double metal layer in the vessel wall, which is linked to delayed healing. Furthermore there might be a higher risk of malapposition of both struts of the bare metal and the newly implanted drug-eluting stents. These phenomenon's might give rise to an increased risk of stent thrombosis in this patient population. Recently, drug-eluting balloons (DEB) were proposed as a new treatment strategy for bare metal stent restenosis. The initial results of this technique look promising.

Aim: To compare healing processes after treatment of BMS ISR with balloon dilatation using DEB versus implantation of DES.

Methods: 50 patients with BMS restenosis (SVG and bifurcation lesions will be excluded) will be randomized into two treatment groups: SeQuent Please drug-eluting balloon dilatation (group I) versus implantation of an everolimus-eluting Xience V stent (group II). At 9 months, a control angiography with OCT pullback of the treated segment is planned.

ELIGIBILITY:
Inclusion Criteria:

1. Patient older than 18 years
2. written informed consent available
3. patient eligible for percutaneous coronary intervention
4. patients with a single or multiple re-stenotic lesion(s) in a previously stented area of a coronary artery (irrelevant whether BMS or DES)
5. Target reference vessel diameter measured by QCA: 2-4 mm
6. Target lesion length measured by QCA < 24 mm
7. Target lesion stenosis measured by QCA: > 70%- < 100%
8. Patients willing to provide written informed consent prior to participation and willing and able to participate in all follow-up evaluations.

Exclusion Criteria:

1. Left ventricular ejection fraction of < 30%
2. Impaired renal function (serum creatinine > 2.0 mg/dl)
3. Target lesion located in bifurcation
4. Previous and/or planned brachytherapy of target vessel
5. Lesion of the left main trunk > 50%, unprotected
6. Known allergies to antiplatelet, anticoagulation therapy, contrast media, paclitaxel or everolimus
7. Pregnant and/or breast-feeding females or females who intend to become pregnant (pregnancy test required)
8. Patients with a life expectancy of less than one year
9. Patients who intend to have a major surgical intervention within 6 months of enrolment in the study.
10. Patient currently enrolled in other investigational device or drug trial
11. Patient not able or willing to adhere to follow-up visits
12. Patients who previously participated in this study. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-05 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Stent strut coverage and stent strut apposition(assessed with OCT) | 9 months

SECONDARY OUTCOMES:
Lumen Loss (in-stent) at 9 months In-segment Late Lumen Loss at 9 months Cumulative MACE rate at 9 months Stent thrombosis at all follow-ups Target vessel revascularisation (TVR) at 12 months Device success | 9 months, 12 months, yearly until 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tom Adriaenssens, MD, Principal Investigator — UZ Leuven; Walter Desmet, MD, PhD, Study Director — UZ Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Adriaenssens T, Dens J, Ughi G, Bennett J, Dubois C, Sinnaeve P, Wiyono S, Coosemans M, Belmans A, D'hooge J, Vrolix M, Desmet W. Optical coherence tomography study of healing characteristics of paclitaxel-eluting balloons vs. everolimus-eluting stents for in-stent restenosis: the SEDUCE (Safety and Efficacy of a Drug elUting balloon in Coronary artery rEstenosis) randomised clinical trial. EuroIntervention. 2014 Aug;10(4):439-48. doi: 10.4244/EIJV10I4A77. PMID 25138182